CLINICAL TRIAL: NCT01903837
Title: A Phase 2, Randomized, Multicenter, Safety, Tolerability, and Dose-Ranging Study of Samidorphan, a Component of ALKS 3831, in Adults With Schizophrenia Treated With Olanzapine
Brief Title: A Study of ALKS 3831 in Adults With Schizophrenia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK3831-302
Record Dates: First submitted 2013-07-05; First posted 2013-07-19 (Estimated); Results first posted 2021-09-08 (Actual); Last update posted 2021-10-06 (Actual); Status verified 2021-09

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Olanzapine; Samidorphan; Alkermes
MeSH Terms: conditions — Schizophrenia | interventions — 3-carboxamido-4-hydroxynaltrexone; Olanzapine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low Dose (Experimental): Olanzapine + low dose samidorphan tablets taken once daily
  Interventions: Drug: Samidorphan (Low Dose); Drug: Olanzapine
- Medium Dose (Experimental): Olanzapine + medium dose samidorphan tablets taken once daily
  Interventions: Drug: Samidorphan (Medium Dose); Drug: Olanzapine
- High Dose (Experimental): Olanzapine + high dose samidorphan tablets taken once daily
  Interventions: Drug: Samidorphan (High Dose); Drug: Olanzapine
- Placebo (Placebo Comparator): Olanzapine + placebo tablets taken once daily
  Interventions: Drug: Placebo; Drug: Olanzapine

INTERVENTIONS:
Drug: Samidorphan (Low Dose) — Tablets taken once daily
  Other Names: Low dose samidorphan (ALKS 33)
  Arms: Low Dose
Drug: Samidorphan (Medium Dose) — Tablets taken once daily
  Other Names: Medium dose samidorphan (ALKS 33)
  Arms: Medium Dose
Drug: Samidorphan (High Dose) — Tablets taken once daily
  Other Names: High dose samidorphan (ALKS 33)
  Arms: High Dose
Drug: Placebo — Tablets taken once daily
  Arms: Placebo
Drug: Olanzapine — Tablets taken once daily

SUMMARY:
This is a Phase 2, randomized, placebo-controlled multicenter study, which will be conducted in 2 parts. The study duration for each subject will be approximately 33 weeks and will include 25 study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 50 years, inclusive
* Body mass index (BMI) of 17-30 kg/m2, inclusive
* Diagnosis of schizophrenia that is clinically stable

Exclusion Criteria:

* Initiated 1st antipsychotic treatment within the past 12 months and/or has had symptoms lasting <2 years
* Current diagnosis of alcohol or drug use disorder, moderate or severe
* Clinically significant or unstable medical illness, condition, or disorder
* Pregnant or breastfeeding
* Significant changes in diet or exercise regimen or plans to join a weight management program during the study
* Opioid medications taken within 14 days and/or need to take opioid medication during the study period
* History of hypersensitivity to or intolerance of olanzapine
* Use of olanzapine, clozapine, mesoridazine, chlorpromazine, or thioridazine for more than 1 week during the past year

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 347 (Actual)
Dates: Start 2013-06; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.
Locations (57):
- United States (46):
  - Alkermes Investigational Site, Little Rock, Arkansas
  - Alkermes Investigational Site, Anaheim, California
  - Alkermes Investigational Site, Costa Mesa, California
  - Alkermes Investigational Site, Culver City, California
  - Alkermes Investigational Site, Escondido, California
  - Alkermes Investigational Site, Garden Grove, California
  - Alkermes Investigational Site, National City, California
  - Alkermes Investigational Site, Oakland, California
  - Alkermes Investigational Site, Oceanside, California
  - Alkermes Investigational Site, Orange, California
  - Alkermes Investigational Site, Pico Rivera, California
  - Alkermes Investigational Site, San Diego, California
  - Alkermes Investigational Site, Torrance, California
  - Alkermes Investigational Site, New Britain, Connecticut
  - Alkermes Investigational Site, Washington D.C., District of Columbia
  - Alkermes Investigational Site, Bradenton, Florida
  - Alkermes Investigational Site, Fort Lauderdale, Florida
  - Alkermes Investigational Site, Gainesville, Florida
  - Alkermes Investigational Site, Kissimmee, Florida
  - Alkermes Investigational Site, Leesburg, Florida
  - Alkermes Investigational Site, Oakland Park, Florida
  - Alkermes Investigational Site, Orlando, Florida
  - Alkermes Investigational Site, Atlanta, Georgia
  - Alkermes Investigational Site, Decatur, Georgia
  - Alkermes Investigational Site, Chicago, Illinois
  - Alkermes Investigational Site, Lake Charles, Louisiana
  - Alkermes Investigational Site, Shreveport, Louisiana
  - Alkermes Investigational Site, Rockville, Maryland
  - Alkermes Investigational Site, Flowood, Mississippi
  - Alkermes Investigational Site, Creve Coeur, Missouri
  - Alkermes Investigational Site, St Louis, Missouri
  - Alkermes Investigational Site, Marlton, New Jersey
  - Alkermes Investigational Site, Neptune City, New Jersey
  - Alkermes Investigational Site, Canton, Ohio
  - Alkermes Investigational Site, Mason, Ohio
  - Alkermes Investigational Site, Oklahoma City, Oklahoma
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigational Site, Charleston, South Carolina
  - Alkermes Investigational Site, Memphis, Tennessee
  - Alkermes Investigational Site, Austin, Texas
  - Alkermes Investigational Site, Dallas, Texas
  - Alkermes Investigational Site, DeSoto, Texas
  - Alkermes Investigational Site, Houston, Texas
  - Alkermes Investigational Site, Salt Lake City, Utah
  - Alkermes Investigational Site, Bellevue, Washington
  - Alkermes Investigational Site, Richland, Washington
- Bulgaria (9):
  - Alkermes Investigational Site, Burgas
  - Alkermes Investigational Site, Kazanlak
  - Alkermes Investigational Site, Lovech
  - Alkermes Investigational Site, Novi Iskar
  - Alkermes Investigational Site, Pazardzhik
  - Alkermes Investigational Site, Sofia
  - Alkermes Investigational Site, Tserova Koria
  - Alkermes Investigational Site, Varna
  - Alkermes Investigational Site, Vratsa
- Czechia (2):
  - Alkermes Investigational Site, Brno-mesto
  - Alkermes Investigational Site, Prague

REFERENCES:
- [Result] Martin WF, Correll CU, Weiden PJ, Jiang Y, Pathak S, DiPetrillo L, Silverman BL, Ehrich EW. Mitigation of Olanzapine-Induced Weight Gain With Samidorphan, an Opioid Antagonist: A Randomized Double-Blind Phase 2 Study in Patients With Schizophrenia. Am J Psychiatry. 2019 Jun 1;176(6):457-467. doi: 10.1176/appi.ajp.2018.18030280. Epub 2019 Mar 8. PMID 30845818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included subjects who had a diagnosis of schizophrenia and who had not been exposed to olanzapine, clozapine, mesoridazine, chlorpromazine, or thioridazine for more than 1 week within the previous year or at any time in the 3 months prior to screening. Subjects were enrolled in study sites located in 3 countries: United States, Bulgaria, and the Czech Republic.
Pre-assignment Details: Subjects completed a seven-day lead-in period on open-label olanzapine before being randomized into the 12-week double-blind treatment period. Baseline data includes subjects who completed the lead-in period and were randomized to a treatment group. A total of 347 subjects were enrolled in the study; 309 subjects completed the 1-week olanzapine lead-in period and were randomized to one of the 4 treatment groups in Part A
Groups:
- Olz + Placebo/ Olz+Sam 20mg: Part A: Olanzapine (dose level determined by Investigator) + placebo tablets taken once daily
  Part B: Olanzapine (dose level determined by Investigator) + 20mg Samidorphan tablets taken once daily
  Subjects were transitioned from placebo in Part A to 20mg Samidorphan in Part B
- Olz + Sam 5mg / Olz + Sam 5mg: Part A: Olanzapine (dose level determined by Investigator) + 5mg samidorphan tablets taken once daily
  Part B: Olanzapine (dose level determined by Investigator) + 5mg samidorphan tablets taken once daily
- Olz + Sam 10mg /Olz + Sam 10mg: Part A: Olanzapine (dose level determined by Investigator) + 10mg Samidorphan tablets taken once daily
  Part B: Olanzapine (dose level determined by Investigator) + 10mg Samidorphan tablets taken once daily
- Olz + Sam 20mg/ Olz + Sam 20mg: Part A: Olanzapine (dose level determined by Investigator) + 20mg samidorphan tablets taken once daily
  Part B: Olanzapine (dose level determined by Investigator) + 20mg samidorphan tablets taken once daily
Period: Part A
Arm/Group | Olz + Placebo/ Olz+Sam 20mg | Olz + Sam 5mg / Olz + Sam 5mg | Olz + Sam 10mg /Olz + Sam 10mg | Olz + Sam 20mg/ Olz + Sam 20mg
Started | 75 | 80 | 86 | 68
Completed | 56 | 52 | 58 | 55
Not Completed | 19 | 28 | 28 | 13
Not completed — Withdrawal by Subject | 4 | 9 | 8 | 5
Not completed — Adverse Event | 3 | 6 | 9 | 6
Not completed — Lost to Follow-up | 9 | 7 | 7 | 2
Not completed — Non-compliance with study drug | 1 | 4 | 4 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 1 | 0 | 0
Period: Part B
Arm/Group | Olz + Placebo/ Olz+Sam 20mg | Olz + Sam 5mg / Olz + Sam 5mg | Olz + Sam 10mg /Olz + Sam 10mg | Olz + Sam 20mg/ Olz + Sam 20mg
Started (The number of subjects starting the period is not consistent with the number completing the preceding period. It is expected the number of subjects starting the subsequent period will be the same as the number completing the preceding period. This is because 3 subjects discontinued the study after completing Part A, and did not participate in Part B.) | 54 | 52 | 57 | 55
Completed | 45 | 46 | 52 | 44
Not Completed | 9 | 6 | 5 | 11
Not completed — Lost to Follow-up | 0 | 3 | 3 | 4
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 3
Not completed — Adverse Event | 3 | 0 | 2 | 0
Not completed — Non-compliance with study drug | 2 | 0 | 0 | 1
Not completed — Incarceration | 2 | 0 | 0 | 1
Not completed — Physician Decision | 1 | 0 | 0 | 2
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Olz + Placebo: Olanzapine (dose level determined by Investigator) and placebo tablets taken once daily
- Olz + Sam 5mg: Olanzapine (dose level determined by Investigator) and 5mg Samidorphan tablets taken once daily
- Olz + Sam 10mg: Olanzapine (dose level determined by Investigator) and 10mg Samidorphan tablets taken once daily
- Olz + Sam 20mg: Olanzapine (dose level determined by Investigator) and 20mg Samidorphan tablets taken once daily
- Total: Total of all reporting groups
Arm/Group | Olz + Placebo | Olz + Sam 5mg | Olz + Sam 10mg | Olz + Sam 20mg | Total
Number analyzed (Participants) | 75 | 80 | 86 | 68 | 309
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (8.14) | 37.9 (8.62) | 38.1 (8.00) | 39.3 (8.38) | 38.8 (8.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 20 | 21 | 18 | 81
  Male | 53 | 60 | 65 | 50 | 228
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 5 | 5 | 3 | 17
  Not Hispanic or Latino | 71 | 75 | 81 | 65 | 292
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 1 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 1 | 3
  Black or African American | 44 | 53 | 50 | 42 | 189
  White | 28 | 26 | 35 | 23 | 112
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 60 | 68 | 70 | 60 | 258
  Czechia | 0 | 0 | 1 | 0 | 1
  Bulgaria | 15 | 12 | 15 | 8 | 50
Height [Mean (Standard Deviation); unit: centimeters] | 173.4 (8.07) | 173.5 (10.76) | 174.8 (10.27) | 174.1 (9.99) | 174 (9.82)
Weight [Mean (Standard Deviation); unit: kilograms] | 75.6 (12.30) | 77.5 (13.07) | 76.7 (13.67) | 75.4 (12.81) | 76.4 (12.96)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms/meters^2] | 25.1 (3.40) | 25.7 (3.18) | 25.0 (3.23) | 24.8 (3.41) | 25.2 (3.30)
Body Mass Index (BMI) Group [Count of Participants; unit: Participants]
  Underweight (<18.5) | 1 | 0 | 1 | 1 | 3
  Normal (18.5 to <25) | 32 | 31 | 42 | 32 | 137
  Overweight (25 to <30) | 42 | 46 | 43 | 34 | 165
  Obese (>=30) | 0 | 3 | 0 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Total Positive and Negative Syndrome Scale (PANSS) Score
Description: Change from baseline (Day 8) to Day 92 (end of study Part A).
  The PANSS is a 30-item scale measuring severity of schizophrenia symptoms. Symptom severity for each item is rated on a 7-point scale (1 = absent; 7 = extreme), and the total score is added together, with a minimum score of 30 and a maximum score of 210. A higher score indicates more severe symptoms, while a lower score indicates less severe symptoms.
Time Frame: Baseline (Day 8) to Day 92 (end of study Part A)
Population: Full Analysis Set (FAS) 1 efficacy analysis population included all randomized subjects who received at least one dose of study drug and had at least one postbaseline assessment of Positive and Negative Syndrome Scale (PANSS) total score.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Part A FAS 1 - Olz + Placebo: Subjects who were randomized to olanzapine + placebo in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1 - Olz + Sam 5mg: Subjects who were randomized to olanzapine + samidorphan 5mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz+ Sam 10mg: Subjects who were randomized to olanzapine + samidorphan 10mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz+ Sam 20mg: Subjects who were randomized to olanzapine + samidorphan 20mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
Arm/Group | Part A FAS 1 - Olz + Placebo | Part A FAS 1 - Olz + Sam 5mg | Part A FAS 1- Olz+ Sam 10mg | Part A FAS 1- Olz+ Sam 20mg
Number analyzed (Participants) | 74 | 75 | 83 | 68
units on a scale | -2.9 (0.82) | -1.5 (0.85) | -2.7 (0.79) | -2.5 (0.83)
Statistical Analysis 1: Comparison: Part A FAS 1 - Olz + Placebo vs Part A FAS 1 - Olz + Sam 5mg vs Part A FAS 1- Olz+ Sam 10mg vs Part A FAS 1- Olz+ Sam 20mg; Test type: Equivalence — Equivalence margin of 10 points; p = 0.3, Least Square Mean Difference; Least Square Mean Difference = 0.3, 95% CI 2-sided [-2.0 to 2.6], Standard Error of Mean 1.17

2. Secondary Outcome: Percent Change in Body Weight (Kilogram) From Baseline to Day 92
Description: Percent change from baseline (Day 8) to the end of Part A (Day 92)
Time Frame: Baseline (Day 8) to Day 92 (end of study Part A)
Population: Full Analysis Set (FAS) 1 efficacy analysis population included all randomized subjects who received at least one dose of study drug and had at least one postbaseline assessment of Positive and Negative Syndrome Scale (PANSS) total score. FAS 2 efficacy analysis population included all FAS 1 subjects who gained weight during the 1-week OLZ lead-in period prior to randomization and had at least one postbaseline weight assessment.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent change
Groups:
- Part A FAS 1- Olz + Sam 10mg: Subjects who were randomized to olanzapine + samidorphan 10mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz + Sam 20mg: Subjects who were randomized to olanzapine + samidorphan 20mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 2- Olz + Placebo: All FAS 1 subjects who were randomized to olanzapine + placebo in study Part A, gained weight during the first week of olanzapine treatment prior to randomization, and had at least one post-baseline weight assessment.
- Part A FAS 2- Olz + Sam 5mg: All FAS 1 subjects who were randomized to olanzapine + samidorphan 5mg in study Part A, gained weight during the first week of olanzapine treatment prior to randomization, and had at least one post-baseline weight assessment.
- Part A FAS 2- Olz + Sam 10mg: All FAS 1 subjects who were randomized to olanzapine + samidorphan 10mg in study Part A, gained weight during the first week of olanzapine treatment prior to randomization, and had at least one post-baseline weight assessment.
- Part A FAS 2- Olz + 20mg: All FAS 1 subjects who were randomized to olanzapine + samidorphan 20mg in study Part A, gained weight during the first week of olanzapine treatment prior to randomization, and had at least one post-baseline weight assessment.
Arm/Group | Part A FAS 1 - Olz + Placebo | Part A FAS 1 - Olz + Sam 5mg | Part A FAS 1- Olz + Sam 10mg | Part A FAS 1- Olz + Sam 20mg | Part A FAS 2- Olz + Placebo | Part A FAS 2- Olz + Sam 5mg | Part A FAS 2- Olz + Sam 10mg | Part A FAS 2- Olz + 20mg
Number analyzed (Participants) | 74 | 75 | 83 | 67 | 45 | 50 | 53 | 46
percent change | 4.1 [3.2 to 5.0] | 2.8 [1.8 to 3.7] | 2.1 [1.3 to 3.0] | 2.9 [1.9 to 3.8] | 5.3 [4.2 to 6.4] | 3.8 [2.7 to 4.9] | 2.2 [1.2 to 3.3] | 1.6 [0.5 to 2.7]
Statistical Analysis 1: Comparison: Part A FAS 1 - Olz + Placebo vs Part A FAS 1 - Olz + Sam 5mg vs Part A FAS 1- Olz + Sam 10mg vs Part A FAS 1- Olz + Sam 20mg; Test type: Superiority; p = 0.006, Mixed Models Analysis
Statistical Analysis 2: Comparison: Part A FAS 2- Olz + Placebo vs Part A FAS 2- Olz + Sam 5mg vs Part A FAS 2- Olz + Sam 10mg vs Part A FAS 2- Olz + 20mg; Test type: Superiority; p < 0.001, Mixed Models Analysis

3. Secondary Outcome: Absolute Change in Body Weight (kg) From Baseline to Day 92
Description: Change from randomization (Day 8) to the end of Part A (Week 12; Day 92)
Time Frame: Baseline (Day 8) to Day 92 (end of study Part A)
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: kg
Groups:
- Part A FAS 1- Olz + Placebo: Subjects who were randomized to olanzapine + placebo in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz + Sam 5mg: Subjects who were randomized to olanzapine + 5mg samidorphan in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz + Sam 10mg: Subjects who were randomized to olanzapine + 10mg samidorphan in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 1- Olz + Sam 20mg: Subjects who were randomized to olanzapine + 20mg samidorphan in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 2- Olz + Sam 20mg: All FAS 1 subjects who were randomized to olanzapine + samidorphan 20mg in study Part A, gained weight during the first week of olanzapine treatment prior to randomization, and had at least one post-baseline weight assessment.
Arm/Group | Part A FAS 1- Olz + Placebo | Part A FAS 1- Olz + Sam 5mg | Part A FAS 1- Olz + Sam 10mg | Part A FAS 1- Olz + Sam 20mg | Part A FAS 2- Olz + Placebo | Part A FAS 2- Olz + Sam 5mg | Part A FAS 2- Olz + Sam 10mg | Part A FAS 2- Olz + Sam 20mg
Number analyzed (Participants) | 74 | 75 | 83 | 67 | 45 | 50 | 53 | 47
kg | 2.9 [2.2 to 3.6] | 2.1 [1.4 to 2.8] | 1.5 [0.9 to 2.2] | 2.2 [1.5 to 2.9] | 3.8 [2.9 to 4.6] | 2.9 [2.1 to 3.7] | 1.5 [0.7 to 2.3] | 1.2 [0.4 to 2.1]
Statistical Analysis 1: Comparison: Part A FAS 1- Olz + Placebo vs Part A FAS 1- Olz + Sam 5mg vs Part A FAS 1- Olz + Sam 10mg vs Part A FAS 1- Olz + Sam 20mg; Test type: Superiority; p = 0.018, Mixed Models Analysis
Statistical Analysis 2: Comparison: Part A FAS 2- Olz + Placebo vs Part A FAS 2- Olz + Sam 5mg vs Part A FAS 2- Olz + Sam 10mg vs Part A FAS 2- Olz + Sam 20mg; Test type: Superiority; p < 0.001, Mixed Models Analysis

4. Secondary Outcome: Percentage of Subjects Exhibiting Significant Weight Gain at Day 92
Description: Significant weight gain will include a >=5%, >= 7%, or >=10% gain in body weight from baseline (Day 8) to Day 92 (end of study Part A)
Time Frame: Baseline (Day 8) to Day 92 (end of study Part A)
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Part A FAS 1- Olz + Sam 5mg: Subjects who were randomized to olanzapine + samidorphan 5mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 2- Olz + Placebo: All FAS 1 subjects who were randomized to olanzapine + placebo in study Part A, gained weight during the first week of olanzapine treatment prior to randomization and had at least one post-baseline weight assessment.
- Part A FAS 2- Olz + Sam 5mg: All FAS 1 subjects who were randomized to olanzapine + samidorphan 5mg in study Part A, gained weight during the first week of olanzapine treatment prior to randomization and had at least one post-baseline weight assessment.
- Part A FAS 2- Olz + Sam 10mg: Subjects who were randomized to olanzapine + samidorphan 10mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
- Part A FAS 2- Olz + Sam 20mg: Subjects who were randomized to olanzapine + samidorphan 20mg in study Part A, received at least one dose of study drug, and had at least one post-baseline assessment of PANSS total score
Arm/Group | Part A FAS 1- Olz + Placebo | Part A FAS 1- Olz + Sam 5mg | Part A FAS 1- Olz + Sam 10mg | Part A FAS 1- Olz + Sam 20mg | Part A FAS 2- Olz + Placebo | Part A FAS 2- Olz + Sam 5mg | Part A FAS 2- Olz + Sam 10mg | Part A FAS 2- Olz + Sam 20mg
Number analyzed (Participants) | 56 | 52 | 59 | 54 | 35 | 35 | 36 | 35
Participants
  >= 5% weight gain | 20 | 18 | 16 | 16 | 14 | 13 | 8 | 8
  >= 7% weight gain | 14 | 8 | 9 | 12 | 11 | 7 | 4 | 7
  >=10% weight gain | 10 | 3 | 4 | 5 | 8 | 3 | 3 | 1

5. Secondary Outcome: Change in Clinical Global Impressions - Severity (CGI-S) From Baseline to Day 92
Description: Change in CGI-S score from baseline (Day 8) to the end of Part A (Week 12; Day 92).
  The CGI-S is a 7-point scale intended to measure the severity of a patient's illness at the time of assessment. Scores range from 1 (normal) to 7(extremely ill), so a higher score is correlative to more severe illness.
Time Frame: Baseline (Day 8) to Day 92 (end of study Part A)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Part A FAS 1 - OLZ + Placebo | Part A FAS 1 - Olz + Sam 5mg | Part A FAS 1- Olz + Sam 10mg | Part A FAS 1- Olz + Sam 20mg
Number analyzed (Participants) | 74 | 75 | 83 | 68
units on a scale | -0.0 (0.05) | -0.1 (0.05) | -0.0 (0.05) | -0.1 (0.05)

ADVERSE EVENTS:
Time Frame: Safety assessments are presented for all dosing groups in both Study Parts A and B, i.e. 24 weeks
Groups:
- Part A- Olz + Placebo: Olanzapine (dose level determined by Investigator) + placebo tablets taken once daily
- Part A-Olz + Sam 5mg; Part B- Olz + Sam 5mg / Olz +Sam 5mg: Olanzapine (dose level determined by Investigator) + 5mg samidorphan tablets taken once daily
- Part A- Olz + Sam 10mg; Part B- Olz + Sam 10mg/ Olz + Sam 10mg: Olanzapine (dose level determined by Investigator) + 10mg Samidorphan tablets taken once daily
- Part A- Olz + Sam 20mg; Part B-Olz + Sam 20mg/ Olz + Sam 20mg: Olanzapine (dose level determined by Investigator) + 20mg samidorphan tablets taken once daily
- Part B-Olz +Placebo/ Olz+Sam 20mg: Olanzapine (dose level determined by Investigator) + 20mg Samidorphan tablets taken once daily
  Subjects were transitioned from placebo in Part A to 20mg Samidorphan in Part B
Arm/Group | Part A- Olz + Placebo | Part A-Olz + Sam 5mg | Part A- Olz + Sam 10mg | Part A- Olz + Sam 20mg | Part B-Olz +Placebo/ Olz+Sam 20mg | Part B- Olz + Sam 5mg / Olz +Sam 5mg | Part B- Olz + Sam 10mg/ Olz + Sam 10mg | Part B-Olz + Sam 20mg/ Olz + Sam 20mg
All-Cause Mortality (participants affected / at risk) | 0/75 | 0/80 | 0/86 | 0/68 | 0/54 | 0/52 | 0/57 | 0/55
Serious Adverse Events (participants affected / at risk) | 2/75 | 3/80 | 4/86 | 4/68 | 1/54 | 1/52 | 1/57 | 0/55
Other Adverse Events (participants affected / at risk) | 33/75 | 25/80 | 33/86 | 33/68 | 11/54 | 10/52 | 11/57 | 12/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A- Olz + Placebo (N=75) | Part A-Olz + Sam 5mg (N=80) | Part A- Olz + Sam 10mg (N=86) | Part A- Olz + Sam 20mg (N=68) | Part B-Olz +Placebo/ Olz+Sam 20mg (N=54) | Part B- Olz + Sam 5mg / Olz +Sam 5mg (N=52) | Part B- Olz + Sam 10mg/ Olz + Sam 10mg (N=57) | Part B-Olz + Sam 20mg/ Olz + Sam 20mg (N=55)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Schizophrenia (Psychiatric disorders) | 1 | 2 | 1 | 3 | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part A- Olz + Placebo (N=75) | Part A-Olz + Sam 5mg (N=80) | Part A- Olz + Sam 10mg (N=86) | Part A- Olz + Sam 20mg (N=68) | Part B-Olz +Placebo/ Olz+Sam 20mg (N=54) | Part B- Olz + Sam 5mg / Olz +Sam 5mg (N=52) | Part B- Olz + Sam 10mg/ Olz + Sam 10mg (N=57) | Part B-Olz + Sam 20mg/ Olz + Sam 20mg (N=55)
Weight increased (Investigations) | 9 | 8 | 9 | 6 | 3 | 6 | 2 | 3
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Somnolence (Nervous system disorders) | 3 | 10 | 11 | 8 | 2 | 0 | 3 | 4
Sedation (Nervous system disorders) | 3 | 0 | 4 | 8 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 3 | 6 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 4 | 3 | 1 | 1 | 1 | 0 | 4 | 1
Tremor (Nervous system disorders) | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 2 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 5 | 4 | 5 | 6 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 4 | 2 | 5 | 6 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 5 | 2 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 6 | 0 | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 6 | 5 | 5 | 6 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 4 | 2
Toothache (Gastrointestinal disorders) | 4 | 0 | 0 | 2 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should an Investigator desire to disclose study results, Sponsor will review the results disclosure prior to public release and can embargo the disclosure for a period of at least 60 days. Revisions to the disclosure will be negotiated in good faith. For a multicenter study the Investigators agree to publish/publicly present the results together with the other sites for the 12 month period after study results are available unless Sponsor grants written permission in advance.

DOCUMENTS (2):
  • Study Protocol (2014-06-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT01903837/Prot_000.pdf
  • Statistical Analysis Plan (2014-12-02): https://cdn.clinicaltrials.gov/large-docs/37/NCT01903837/SAP_001.pdf